CLINICAL TRIAL: NCT01966042
Title: Phase II Study of Intramyocardial Injection of Autologous Bone Marrow Stem Cells for Refractory Angina in Patients With Normal or Slightly Reduced Left Ventricular Function.
Brief Title: Study Protocol of Intramyocardial Injection of Autologous Bone Marrow Stem Cells for Refractory Angina
Acronym: ReACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CellPraxis Bioengenharia Ltda. (Industry)
Collaborators: Cryopraxis Criobiologia Ltda. (Industry); Federal University of São Paulo (Other); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cell 0314/05; 0314/05 (Other: CEP)
Record Dates: First submitted 2013-10-14; First posted 2013-10-21 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Refractory Angina
Keywords: Refractory angina; Cell Therapy; Bone Marrow; Mononuclear Cells
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Therapy (Experimental): All subjects enrolled in the study underwent:
  Local Sedation; Bone Marrow Aspiration; Minithoracotomy; Autologous bone marrow mononuclear cells infusion.
  Interventions: Procedure: Local sedation; Procedure: Bone Marrow Aspiration; Procedure: Minithoracotomy; Biological: Autologous bone marrow mononuclear cells infusion

INTERVENTIONS:
Procedure: Local sedation — All subjects enrolled in the study underwent local sedation for bone marrow aspiration.
Procedure: Bone Marrow Aspiration — All subjects enrolled in the study underwent bone marrow aspiration after they had been anesthetized from the posterior iliac crest. The sample was aspirated into a series of sterile syringes and brought to the cell processing room/laboratory. The processing was in accordance to the Standard Operating Procedure developed observing Good Practice Guidelines.
Procedure: Minithoracotomy — The surgical procedure used as cardiac access route was the left anterolateral thoracotomy or left anterior minithoracotomy, depending on the segment of the left ventricle to be treated, allowing the good access to the viable myocardial areas.
Biological: Autologous bone marrow mononuclear cells infusion — Once the subject had his or her chest opened and the coronary anatomy reviewed by examination of the pre-operatory nuclear scan to define the area of ischemia, the surgeon drew up the cells into a series of syringes and injected the entire contents of the cell preparation in a series of injections directly into the myocardium.

SUMMARY:
Therapeutic neovascularization is an innovative strategy for cardiac tissue recovery due to chronic, intense ischemia. Thus stem cell therapy has become a promising procedure for the large number of patients with refractory angina due to coronary disease, despite of the use of multiple anti-angina medications, remain severely symptomatic with disabling angina.

Stem cell therapy using autologous cells from the patient's bone marrow, has been shown to be safe and associated with improved myocardial perfusion, reducing the symptoms of advanced coronary artery disease and increasing the functional capacity of patients whose therapeutic armamentarium available today has been exhausted.

The study hypothesis was that the infusion of autologous mononuclear cells derived from the patient's bone marrow and delivered via intramyocardial injection in patients with refractory angina and normal or slightly depressed ventricular function, promote improvement in the anginal symptoms and myocardial perfusion by the inducing neoangiogenesis.

DETAILED DESCRIPTION:
This was a phase II, non-controlled (single arm) and open label clinical trial. The study was approved by the Institutional Review Board (IRB) and all patients gave informed consent prior to participation.

Refractory angina patients were defined as those with functional class IV (angina at rest) according to the Canadian Cardiovascular Society Angina Classification (CCSAC) despite maximum medical therapy, not suitable for conventional myocardial revascularization and viable myocardium confirmed by nuclear imaging.

Patients were evaluated according to different parameters, for a total period of 12 months, and the primary objectives were:

1. Improvement in functional class and angina symptoms (CCSAC) of the patients with refractory angina pectoris after the infusion of autologous bone marrow mononuclear cells after the intervention;
2. Improvement in myocardial perfusion before and after cell delivery;
3. Evaluate the safety of the delivery of autologous bone marrow mononuclear cells route in individuals with refractory angina.

In the screening evaluation, individuals with the presumptive diagnosis of class IV refractory angina and who met all study criteria were approached about the possibility of participating in the study by the principal investigator. Then, the patients were submitted to a baseline evaluation with a serious of blood and image tests.

The interventions were the Bone Marrow Aspiration - For each patient, a total of 100 cc of bone marrow was aspirated from the iliac crest at the time of anesthesia for their cardiac surgery - and the Infusion - After processing the cells, the surgeon delivered it by a series of epicardial injections into the left ventricular myocardium.

The processing of bone marrow autologous cells aimed to enrich the content of the bone marrow aspirate, separating the mononuclear fraction from the cells which were already differentiated.

The postoperative stage was conducted in an identical way to that of patients who undergo to a myocardial revascularization surgery. It is important to mention that both the ICU and the ward time varied according to the patient's individual evolution.

Finally, the first follow up visit took place at 1 month after the surgery. The subsequent visits were held at 3, 6 and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 21 years old;
* Documented coronary artery disease by angiography and confirmed ischemia by myocardial perfusion scintigraphy with physical or pharmacological stress;
* Class IV angina pectoris (CCSAC) that is unresponsive to optimized dose of at least two anti-anginal medications including nitrates, beta blocker, calcium channel blocker or Ranolazine) as well as aspirin or other anti-platelet agent plus statin therapy;
* Considered to not be a candidate for either percutaneous catheter or surgical myocardial revascularization due to either anatomical type, extent of coronary disease in the target vessel, or caliber of the distal vessels;
* Ejection fraction of > 45% by Transthoracic echocardiogram with Doppler by the Simpson method;
* Myocardial perfusion scintigraphy showing that the areas of myocardial ischemia supply viable tissue.

Exclusion Criteria:

* Significant Valvular Heart Disease;
* Chronic kidney disease requiring renal replacement therapy;
* Severe comorbidities associated with the reduction of life expectancy in less than 5 years;
* Ongoing abusive use of alcohol or illegal drugs (Based on the Diagnostic and Statistical Manual (DSM) IV - CAGE questionnaire);
* Positive Serologic test for HIV, Human T-cell lymphotrophic virus (HTLV), Hepatitis A, B and C;
* History of Malignant neoplasia in the last 2 years;
* Participation into other studies of cell therapy in the last year;
* Pregnancy or Breast-feeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-07; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson A Hossne Junior, MD, PhD, Principal Investigator — Federal University of São Paulo; Enio Buffolo, MD, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Refractory angina patients routinely undergoing treatment at the São Paulo Hospital, in São Paulo, Brazil, a referral tertiary Federal University Hospital for coronary heart disease, were included in the study. The study protocol (ReACT™) was approved by the local and national ethical committee and all patients provided written informed consent.
Pre-assignment Details: Refractory angina patients were defined as those with functional class IV (angina at rest) according to the Canadian Cardiovascular Society Angina Classification (CCSAC) despite maximum medical therapy, not suitable for conventional myocardial revascularization and with viable myocardium identification.
Groups:
- Cell Therapy: All subjects enrolled in the study underwent bone marrow aspiration and autologous bone marrow mononuclear cells infusion.
  Local sedation: All subjects enrolled underwent local sedation for bone marrow aspiration.
  Bone Marrow Aspiration: All subjects enrolled underwent bone marrow aspiration after anesthesia from the posterior iliac crest. The sample was aspirated into sterile syringes and brought to the cell processing laboratory. The processing was in accordance to the Standard Operating Procedure developed observing Good Practice Guidelines.
  Minithoracotomy: The cardiac access route was the left anterolateral thoracotomy or left anterior minithoracotomy, depending on the segment of the left ventricle to be treated.
  Autologous bone marrow mononuclear cells infusion: Once the subject had his or her chest opened, the surgeon drew up the cells into syringes and injected the entire contents of the cell preparation in a series of injections directly into the myocardium.
Period: Overall Study
Arm/Group | Cell Therapy
Started | 13
Completed | 11
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: One patient died from cardiogenic shock due to anterior myocardial infarction after 5 months of follow-up. One patient, after 47.3 months of ReACT's procedure, migrated to CCSAC 4 and met inclusion criteria again. This patient was submitted to a new ReACT's procedure.
Groups:
- Cell Therapy: All subjects enrolled in the study underwent bone marrow aspiration and infusion of autologous bone marrow mononuclear cells.
  Local sedation: All subjects enrolled in the study underwent local sedation for bone marrow aspiration.
  Bone Marrow Aspiration: All subjects enrolled in the study underwent bone marrow aspiration after anesthesia.
  Minithoracotomy: The cardiac access route was the left anterolateral thoracotomy or left anterior minithoracotomy, depending on the segment of the left ventricle to be treated, allowing the good access to the viable myocardial areas.
  Autologous bone marrow mononuclear cells infusion: Once the subject had his or her chest opened and the coronary anatomy reviewed by examination of the pre-operatory nuclear scan to define the area of ischemia, the surgeon drew up the cells into a series of syringes and injected the entire contents of the cell preparation in a series of injections directly into the myocardium.
Arm/Group | Cell Therapy
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Number; unit: participants]
  Brazil | 13

OUTCOME MEASURES:

1. Primary Outcome: Angina Class Variation
Description: It was evaluated in accordance with the percentage of participants that change the functional class of angina according to CCSAC (Canadian Cardiovascular Society Angina Classification - description below), after treatment. The functional class of angina was also analyzed as an ordinal variable and the median of the functional class was calculated before and after the procedure, at the time of interest (3, 6 and 12 months post treatment), in comparison to baseline, ie. value at 3 months minus value at baseline.
  Screening of Functional Graduation of Stable Angina:
  I - Angina only occurs after a fast or prolonged and strenuous effort during work or recreation.
  II - Slight limitation to everyday activities. III - Considerable limitation of common physical activity. IV - Inability to perform any physical activity without discomfort, the symptoms can be present at rest.
Time Frame: 3, 6 and 12 months
Measure: Median (Standard Deviation); unit: Angina Classification
Arm/Group | Cell Therapy
Number analyzed (Participants) | 13
Angina Classification
  Angina Class at 3 Months | -2.0 (1.1)
  Angina Class at 6 Months | -1.0 (1.3)
  Angina Class at 12 Months | -0.5 (0.9)
  Angina Class at Baseline | 4.0 (0.0)
Statistical Analysis 1: Comparison: Cell Therapy; Test type: Superiority or Other; p < 0.001, Friedman test (n=13)

2. Secondary Outcome: Functional Change Evaluation
Description: Analysis of Left Ventricular Ejection Fraction (in %), by echocardiogram.
Time Frame: Baseline and 12 months
Measure: Median (Standard Deviation); unit: percentage of Left Ventrical Ejection
Arm/Group | Cell Therapy
Number analyzed (Participants) | 11
percentage of Left Ventrical Ejection
  LVEF at baseline | 59.2 (8.9)
  LVEF at 12 months | 61.6 (6.3)

3. Other Pre Specified Outcome: Life Quality
Description: Analysis of the variation in life quality questionnaire - Short Form Health Survey (SF-36) was performed. Each domain of the questionnaire was evaluated as a quantitative variable and the medians were retrieved before and after the procedure.
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
  It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  One patient was lost before answering the questionnaire post procedure.
Time Frame: Baseline and 12 months
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Cell Therapy
Number analyzed (Participants) | 10
units on a scale
  Physical Function Pre-procedure | 20.0 (27.1)
  Physical Function Post-procedure | 72.5 (24.5)
  Role-Physical Pre-procedure | 0.0 (31.6)
  Role-Physical Post-procedure | 100.0 (33.7)
  Bodily Pain Pre-procedure | 11.0 (17.3)
  Bodily Pain Post-procedure | 100.0 (35.1)
  General Health Pre-procedure | 20.0 (20.0)
  General Health Post-procedure | 72.0 (19.7)
  Vitality Pre-procedure | 40.0 (22.1)
  Vitality Post-procedure | 95 (31.4)
  Social Function Pre-procedure | 12.5 (30.3)
  Social Function Post-procedure | 100.0 (39.3)
  Role-Emotional Pre-procedure | 100.0 (31.6)
  Emotional Post-procedure | 100.0 (36.0)
  Mental Health Pre-procedure | 70.0 (33.3)
  Mental Health Post-procedure | 98.0 (23.9)

4. Secondary Outcome: Functional Change Evaluation
Description: Analysis of objective improvement in myocardial ischemia (in %), by stress technetium scintigraphy.
Time Frame: Baseline, 6 and 12 months
Measure: Median (Standard Deviation); unit: percentage of area change
Arm/Group | Cell Therapy
Number analyzed (Participants) | 11
percentage of area change
  Myocardium Ischemic Area change after 6 months | -15 (48)
  Myocardium Ischemic Area change after 12 months | -100 (37.1)

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Cell Therapy
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cell Therapy (N=13)
Inferior myocardial infarction (Cardiac disorders) | 1 (1) — The first patient died from inferior myocardial infarction after 5 years of follow-up.
Anterior myocardial infarction (Cardiac disorders) | 1 (1) — One patient died from cardiogenic shock due to anterior myocardial infarction after 5 months of follow-up.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cell Therapy (N=13)
Angina (Cardiac disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to ethical aspects and the inability to justify the use of a surgical intramyocardial placebo in this population, this was non-randomized, open study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less